CLINICAL TRIAL: NCT05289713
Title: A Randomized, Controlled Multicenter Feasibility Pilot Trial on Imaging Confirmed Uncomplicated Acute Appendicitis: Appendectomy vs. Symptomatic Treatment in Pediatric Patients (the APPSYPP) Trial Study Protocol
Brief Title: Appendectomy vs. Symptomatic Treatment in Uncomplicated Acute Appendicitis Among Pediatric Patients
Acronym: APPSYPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Tampere University Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Janne Suominen, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APPSYPP
Record Dates: First submitted 2022-02-08; First posted 2022-03-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Appendicitis
Keywords: uncomplicated acute appendicitis; symptomatic treatment; spontaneous resolution
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): In the surgery group, patients undergo laparoscopic appendectomy within 18 hours after randomization.
  Interventions: Procedure: appendectomy
- Symptomatic treatment (Active Comparator): Symptomatically treated patients are hospitalized for at least 24 hours, and receive intravenous fluids and analgesics according to standard clinical practice.
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Procedure: appendectomy — Laparoscopic appendectomy is performed within 18 hours after randomization in the surgery group. Patients in the symptomatic treatment group are carefully monitored and the same intervention (laparoscopic appendectomy) is performed in case of treatment failure.

SUMMARY:
The APPSYPP trial is a randomized national multicenter feasibility superiority pilot study comparing appendectomy with symptomatic treatment in children with imaging-confirmed uncomplicated acute appendicitis. Patients are recruited from all five Finnish university hospitals. Inclusion criteria are: 1) age 7-15 years, 2) imaging-confirmed uncomplicated acute appendicitis (no appendicolith, perforation, abscess, or tumor suspicion), and 3) CRP ≤ 65 mg/l. Patients are randomized to receive emergency appendectomy or symptomatic treatment. In the surgery group, patients undergo laparoscopic appendectomy within 18 hours after randomization. In order to ensure patient safety, symptomatically treated patients are hospitalized for at least 24 hours, and receive intravenous fluids and analgesics according to standard clinical practice. Primary outcome is treatment success at 30 days defined by not fulfilling any of the treatment failure criteria. In the surgery group, treatment failure is defined as normal appendiceal histopathology or any postintervention complication requiring general anesthesia. In the symptomatic treatment group, treatment failure is defined as inability to discharge from hospital without appendectomy within 48 hours after randomization with a finding of histopathologically inflamed appendix, appendectomy during the initial hospital stay due to clinical progression of appendicitis with histopathologically and surgically confirmed complicated acute appendicitis, appendectomy with a histopathological finding of acute appendicitis after hospital discharge, or any complication of appendicitis requiring general anesthesia. Predefined secondary outcomes include later appendectomies, recurrence of histopathologically confirmed appendicitis and associated symptoms, postintervention complications, return to normal daily activities, quality of, resolution of appendicitis in US imagining after 1 month of symptomatic treatment, comparison of US and MRI findings at presentation, and differences in serum biomarkers and fecal microbiota composition.

DETAILED DESCRIPTION:
While antibiotic treatment is an effective and safe treatment for most adults and children with imaging-confirmed uncomplicated acute appendicitis, emerging evidence further indicates that antibiotics and symptomatic treatment strategies may have similar efficacy and safety in uncomplicated acute appendicitis among adults. There are no randomized studies comparing appendectomy to symptomatic treatment in children.

The APPSYPP trial is a randomized national multicenter feasibility superiority pilot study comparing appendectomy with symptomatic treatment in children with imaging-confirmed uncomplicated acute appendicitis. Patients are recruited from all five Finnish university hospitals. Inclusion criteria are: 1) age 7-15 years, 2) imaging-confirmed uncomplicated acute appendicitis (no appendicolith, perforation, abscess, or tumor suspicion), and 3) CRP ≤ 65 mg/l. Patients are randomized to receive emergency appendectomy or symptomatic treatment. In the surgery group, patients undergo laparoscopic appendectomy within 18 hours after randomization. In order to ensure patient safety, symptomatically treated patients are hospitalized for at least 24 hours, and receive intravenous fluids and analgesics according to standard clinical practice. Primary outcome is treatment success at 30 days defined by not fulfilling any of the treatment failure criteria. In the surgery group, treatment failure is defined as normal appendiceal histopathology or any postintervention complication requiring general anesthesia. In the symptomatic treatment group, treatment failure is defined as inability to discharge from hospital without appendectomy within 48 hours after randomization with a finding of histopathologically inflamed appendix, appendectomy during the initial hospital stay due to clinical progression of appendicitis with histopathologically and surgically confirmed complicated acute appendicitis, appendectomy with a histopathological finding of acute appendicitis after hospital discharge, or any complication of appendicitis requiring general anesthesia.

The APPSYPP feasibility trial aims to assess the symptomatic treatment in children with imaging-confirmed uncomplicated acute appendicitis and whether this can safely be studied in a larger patient cohort in the future.

ELIGIBILITY:
Inclusion Criteria:

* age 7-15 years
* clinical diagnosis of uncomplicated acute appendicitis confirmed by US and/or MRI: adequately visualized appendix with a diameter of 6.1-11.0 mm without evidence of perforation, abscess, appendicolith or tumor suspicion
* CRP ≤ 65 mg/l

Exclusion Criteria:

* inability to give informed consent
* age under 7 or over 15 years
* antibiotic administration within 14 days prior to enrolment
* any previous treatment for acute appendicitis
* severe nausea and/or vomiting preventing oral fluid intake
* systemic disease potentially compromising the safety of symptomatic treatment of acute appendicitis (e.g. type 2 diabetes, malignancy, immune deficiency, or a medical condition requiring immunosuppressant medication)
* diffuse peritonitis or complicated acute appendicitis at imaging (perforation, abscess, appendicolith or tumor suspicion)
* inadequately visualized appendix
* age and sex adjusted BMI over 27 kg/m2 and no MRI performed
* CRP > 65 mg/l.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success at 30d follow-up. | 30 days
  Treatment success is defined by not fulfilling any of the following treatment failure criteria.
  Treatment failure in the surgery group:
  * Normal histopathology of the removed appendix.
  * Any complication of acute appendicitis or surgery requiring general anesthesia (GA) within 30 d.
  Treatment failure in the symptomatic treatment group:
  * Inability to discharge from hospital within 48 h after randomization without appendectomy due to persisting symptoms and unmet discharge criteria with a finding of histopathologically inflamed appendix.
  * Appendectomy due to clinical suspicion of progressive appendicitis including increasing pain not responding to the defined non-opioid analgesics during the initial hospital stay with a finding of histopathologically and surgically confirmed complicated acute appendicitis.
  * Appendectomy with a histopathologically confirmed acute appendicitis after hospital discharge within 30 d.
  * Any complication of AA reiring GA within 30 d.

SECONDARY OUTCOMES:
Postintervention complications | 1 year
  Categorized according to Clavien-Dindo classification (Grades I-V).
Recurrent appendicitis | 1 year
  Recurrence of appendicitis (Histopathological diagnosis).
Recurrent symptoms | 1 year
  The number of emergency department visits or hospitalizations due to symptoms related to appendicitis.
Recovery of normal daily activities | 1 year
  Recovery to normal daily activities, school and sports. Reported in days.
QoL | 1 year
  Quality of life evaluated by PedsQL, a validated questionnaire
Resolution of acute appendicitis | 1 month
  Resolution of acute appendicitis, verified by US imaging.
Comparison of US and MRI in diagnostics | 1 month
  Comparison of US and MRI findings (appendix visibility/normal/uncomplicated/complicated appendicitis) at presentation in the same patient. Percentage (%) of patients with either normal appendix, uncomplicated appendicitis, complicated appendicitis or not visible appendix. Imaging modalities are compared to each other and with histopathological analysis. Whether MRI imaging can improve diagnostics.

OTHER OUTCOMES:
Serum biomarkers and fecal microbiota | 1 month
  Differences in serum biomarkers and fecal microbiota composition between treatment arms as an exploratory endpoint for future research. Serum biomarkers are investigated using proteomics and fecal microbiota composition is analyzed using a phylogenetic microarray. The microarray consists of oligonucleotide probes for the V1 and V6 regions on the 16S ribosomal RNA gene and summarized as abundancies of species-level, genus-level, and phylum-level groups.

CONTACTS AND LOCATIONS:
Overall Officials: Janne Suominen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
All research data will be collected using an online REDCap database. Baseline data collection from all patients presenting with suspected acute appendicitis are collected in emergency department and all relevant data during the treatment and follow up.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years
Access Criteria: Only partipating researchers have access to data.

REFERENCES:
- [Derived] Puputti J, Suominen JS, Luoto T, Hiltunen P, Ripatti L, Nikoskelainen M, Nuutinen S, Sinikumpu JJ, Tahkola E, Porela-Tiihonen S, Hurme S, Salminen P, Pakarinen MP. A randomized, controlled multicenter feasibility pilot trial on imaging confirmed uncomplicated acute appendicitis: Appendectomy vs. symptomatic treatment in pediatric patients (the APPSYPP) trial study protocol. Contemp Clin Trials. 2022 Dec;123:106970. doi: 10.1016/j.cct.2022.106970. Epub 2022 Oct 22. PMID 36280033